CLINICAL TRIAL: NCT05133466
Title: Odour Characteristics of Human Breast Milk of Chinese Mothers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heilongjiang Feihe Dairy Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-FEIHE-BTBU-001
Record Dates: First submitted 2021-10-25; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Breast Milk Collection
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Northern pattern: Mothers recruited from Beijing
- East coastal pattern: Mothers recruited from Wuxi
- South-western pattern: Mothers recruited from Chengdu

SUMMARY:
It is well known that breast milk exerts many positive effects on the general health, growth and development of infants. When breastfeeding is not possible, infant formula is considered to be an effective substitute to satisfy the regular nutritional demand of infants. At present, researchers make every effort to simulate the nutritional status of breast milk but mostly neglect the important role that odour plays in guiding the baby to recognize breast milk, promoting the baby's sucking behavior and food intake. The odour changes of the breast milk are so far mainly related to storage, lactational stage and maternal diet. To understand the odour characteristics of the human breast milk from different regions in China, 90 mothers will be recruited from three Chinese cities: Beijing, Chengdu and Wuxi, representing three typical regions with very different climate characteristics and diet habits. The breast milk samples as well as infant formulas will be analyzed using the identical state of the art separation and identification techniques to identify the odorous compounds, determine their concentrations in the breast milk and infant formula as well as determine their importance in contributing to the total odour of samples. The final objective of this study will be to mimic the odour of the breast milk and to understand the difference of breast milk odour from different regions with very different climate and diet composition, as well as to identify the odour deviation of the infant formula from the breast milk. Our results will provide references for the preparation of new infant formula with both nutritional ingredents and odour characteristics simulating that of breast milk.

ELIGIBILITY:
Inclusion Criteria:

* Lactating mother aged 25 ~ 35 years
* Breastfeeding infants (aged 15 ~180 days) and express sufficient breast milk
* Mother is in good health and has balanced nutrition
* Mother is non smoker and non alcoholic, no smokers living in the same apartment
* Voluntarily signed the Informed Consent Form

Exclusion Criteria:

* Mother or newborn infant has major diseases
* Mother participating in any other nutritional or pharmaceutical intervention studies recently
* Other conditions that are not suitable for this study

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy lactating mothers (aged 25-35 years) who breast-feed their infants (aged 15-180 days).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Odour active compound and their concentrations | Up to 2 years
  Gas chromatography-olfactometry/mass spectrometry and other state of the art equipments and protocols will be employed to identify the odour active compounds in the samples, and their concentration and importance in contributing to the odour will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Health Science Center, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Yu M, Xie Q, Song H, Wang L, Sun H, Jiang S, Zhang Y, Zheng C. Characterization of the odor compounds in human milk by DHS/GC x GC-O-MS: A feasible and efficient method. Food Res Int. 2023 Dec;174(Pt 1):113597. doi: 10.1016/j.foodres.2023.113597. Epub 2023 Oct 21. PMID 37986460